CLINICAL TRIAL: NCT00522379
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, 5-arm, Parallel-group Trial to Assess Rotigotine Transdermal System Dose Response in Subjects With Advanced-stage Parkinson's Disease
Brief Title: Trial to Assess Parkinson's Disease (PD) Symptom Control to Four Doses of Rotigotine in a Transdermal Patch
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP0921
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Results first posted 2012-12-10 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2012-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; rotigotine; patch; transdermal; dopamine agonist; off time; Neupro
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Rotigotine 2 mg/24 hr (Experimental)
  Interventions: Drug: Rotigotine
- Rotigotine 4 mg/24 hr (Experimental)
  Interventions: Drug: Rotigotine
- Rotigotine 6 mg/24 hr (Experimental)
  Interventions: Drug: Rotigotine
- Rotigotine 8 mg/24 hr (Experimental)
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rotigotine — 2 mg/24 hr (one 10 cm^2) transdermal patch applied daily for titration and maintenance period - 16 weeks
  Other Names: Neupro
  Arms: Rotigotine 2 mg/24 hr
Drug: Rotigotine — 4 mg/24 hr (one 20 cm^2) transdermal patch applied daily for titration and maintenance period - 16 weeks
  Other Names: Neupro
  Arms: Rotigotine 4 mg/24 hr
Other: Placebo — Placebo transdermal patch applied daily
  Arms: Placebo
Drug: Rotigotine — 6 mg/24 hr (one 10 cm^2 & one 20 cm^2) transdermal patches applied daily for titration and maintenance period - 16 weeks
  Other Names: Neupro
  Arms: Rotigotine 6 mg/24 hr
Drug: Rotigotine — 8 mg/24 hr (two 10 cm^2 & one 20 cm^2) transdermal patches applied daily for titration and maintenance period - 16 weeks
  Other Names: Neupro
  Arms: Rotigotine 8 mg/24 hr

SUMMARY:
The purpose of this study is to show Rotigotine dose response at four doses of Rotigotine used with L-dopa in treating advanced stage Parkinson's disease.

DETAILED DESCRIPTION:
To maintain treatment blind, two different active patch sizes were used (10 cm^2 & 20 cm^2). Placebo patches matched according to size and appearance. During the trial subjects applied up to three patches, active and placebo, to achieve their assigned daily dose.

ELIGIBILITY:
Inclusion Criteria:

* PD greater than 3 years
* Stable dose L-dopa but symptoms not adequately controlled and have "off" time
* Able and willing to complete diary on specific days

Exclusion Criteria:

* Previous use of rotigotine or Neupro
* Atypical Parkinson's syndrome
* Pallidotomy
* Thalamotomy
* Deep brain stimulation
* Fetal tissue transplant
* Dementia
* Psychosis
* Hallucinations
* Epilepsy
* Renal or hepatic dysfunction
* Clinically relevant cardiac dysfunction
* Symptomatic orthostatic hypotension
* Skin sensitivity to adhesives or unresolved contact dermatitis
* History of chronic alcohol or drug abuse
* Pregnant or of child-bearing potential
* Impulse control disorder

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (77):
- United States (62):
  - Birmingham, Alabama
  - Tuscaloosa, Alabama
  - Gilbert, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Fountain Valley, California
  - Fresno, California
  - Irvine, California
  - La Jolla, California
  - Loma Linda, California
  - Oxnard, California
  - Aurora, Colorado
  - New Haven, Connecticut
  - Boca Raton, Florida
  - Bradenton, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Naples, Florida
  - Ocala, Florida
  - Ormond Beach, Florida
  - Pompano Beach, Florida
  - St. Petersburg, Florida
  - Sunrise, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Suwanee, Georgia
  - Chicago, Illinois
  - Anderson, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Southfield, Michigan
  - Golden Valley, Minnesota
  - St Louis, Missouri
  - Missoula, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Commack, New York
  - New York, New York
  - Rochester, New York
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Columbus, Ohio
  - Toledo, Ohio
  - Greensburg, Pennsylvania
  - Souderton, Pennsylvania
  - Upland, Pennsylvania
  - Memphis, Tennessee
  - Lubbock, Texas
  - San Antonio, Texas
  - Midvale, Utah
  - South Ogden, Utah
  - Alexandria, Virginia
  - Richmond, Virginia
  - Roanoke, Virginia
  - Virginia Beach, Virginia
  - Kirkland, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin
- Santiago, Chile, Chile
- India (10):
  - Hyderbad, Andhra Pradesh
  - Bangalore, Kamataka
  - Mangalore, Kamataka
  - Mysore, Karnataka
  - Calicut, Kerala
  - Thiruvananthapuram, Kerala
  - Indore, Madhya Pradesh
  - Mumbai, Maharashtra
  - Pune, Maharashtra
  - Chennai, Tamil Nadu
- Mexico (2):
  - Aguascalientes, Aguascalientes
  - Monterrey, Nuevo León
- Peru (2):
  - San Isidro, Lima region
  - Santiago de Surco, Lima region

REFERENCES:
- [Derived] LeWitt PA, Poewe W, Elmer LW, Asgharnejad M, Boroojerdi B, Grieger F, Bauer L. The Efficacy Profile of Rotigotine During the Waking Hours in Patients With Advanced Parkinson's Disease: A Post Hoc Analysis. Clin Neuropharmacol. 2016 Mar-Apr;39(2):88-93. doi: 10.1097/WNF.0000000000000133. PMID 26882318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III study started in July 2007 with subjects from the United States, Mexico, Peru, Chile, and India. The primary completion date and study completion date occurred in July 2011.
  The Participant Flow and Baseline Characteristics are represenative of the Safety Set (SS), which is 514 subjects.
Pre-assignment Details: The study outcome measures are representative of the Full Analysis Set (FAS), which is 502 subjects.
  The Full Analysis Set (FAS) consisted of all subjects who were randomized, received at least 1 dose of study medication, and had a valid Baseline primary efficacy measurement and at least 1 valid post-Baseline primary efficacy measurement.
Groups:
- Rotigotine 2 mg/24 hr: 2 mg/24 hr (one 10 cm^2) transdermal patch applied daily for titration and maintenance period - 16 weeks
- Rotigotine 4 mg/24 hr: 4 mg/24 hr (one 20 cm^2) transdermal patch applied daily for titration and maintenance period - 16 weeks
- Rotigotine 6 mg/24 hr: 6 mg/24 hr (one 10 cm^2 & one 20 cm^2) transdermal patches applied daily for titration and maintenance period - 16 weeks
- Rotigotine 8 mg/24 hr: 8 mg/24 hr (two 10 cm^2 & one 20 cm^2) transdermal patches applied daily for titration and maintenance period - 16 weeks
Period: Overall Study
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Started | 101 | 107 | 104 | 94 | 108
Completed | 79 | 84 | 82 | 80 | 81
Not Completed | 22 | 23 | 22 | 14 | 27
Not completed — Adverse Event | 12 | 15 | 12 | 5 | 17
Not completed — Lack of Efficacy | 3 | 0 | 2 | 2 | 7
Not completed — Withdrawal by Subject | 2 | 3 | 1 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 2 | 0 | 0
Not completed — Unsatisfactory Subject Compliance | 1 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 4 | 2 | 2
Not completed — Randomization error | 0 | 0 | 0 | 0 | 1
Not completed — Dispensing error | 1 | 0 | 0 | 1 | 0
Not completed — Subject Moved | 1 | 1 | 0 | 0 | 0
Not completed — Sponsor Request | 0 | 1 | 0 | 0 | 0
Not completed — Family Problem | 0 | 0 | 1 | 0 | 0
Not completed — Site Closed | 0 | 0 | 0 | 1 | 0
Not completed — Subject Withdrawal | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo | Total
Number analyzed (Participants) | 101 | 107 | 104 | 94 | 108 | 514
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 54 | 47 | 49 | 48 | 244
  >=65 years | 55 | 53 | 57 | 45 | 60 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.5) | 64.6 (9.0) | 64.6 (10.4) | 63.2 (11.6) | 64.8 (10.2) | 64.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 31 | 38 | 34 | 155
  Male | 77 | 79 | 73 | 56 | 74 | 359
Region of Enrollment [Number; unit: participants]
  United States | 66 | 72 | 68 | 59 | 69 | 334
  Mexico | 1 | 1 | 2 | 0 | 1 | 5
  Peru | 4 | 3 | 2 | 4 | 3 | 16
  Chile | 2 | 2 | 1 | 2 | 2 | 9
  India | 28 | 29 | 31 | 29 | 33 | 150

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Absolute Time Spent "Off" From Baseline to the End of the Maintenance Period as Recorded by the Subject in a Daily Diary
Description: Time "Off" is defined as when the patient does not have the effect of anti-Parkinson's medication.
Time Frame: From Baseline to the End of the Maintenance Period [16 Weeks Treatment Period (4 weeks Titration Period and 12 weeks Maintenance Period)].
Population: Of the 502 subjects in the Full Analysis Set (FAS), 502 are included in this analysis. The Last Observation Carried Forward (LOCF) method was utilized.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 99 | 103 | 101 | 94 | 105
Hours | -1.948 (2.587) | -2.052 (3.113) | -2.138 (2.721) | -2.360 (2.608) | -1.499 (3.062)

2. Secondary Outcome: The Change in Relative Time Spent "Off" From Baseline to the End of the Maintenance Period as Recorded by the Subject in a Daily Diary
Description: Time "Off" is defined as when the patient does not have the effect of anti-Parkinson's medication.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 99 | 103 | 101 | 94 | 105
Hours | -12.058 (16.517) | -13.463 (20.099) | -13.410 (17.202) | -14.529 (16.531) | -9.250 (18.942)

3. Secondary Outcome: The Change in the Absolute Time Spent "on" From Baseline to the End of the Maintenance Period as Recorded by the Subject in a Daily Diary
Description: Time "On" is defined as when the patient has the effect of anti-Parkinson's medication.
Time Frame: as for outcome 1
Population: Of the 502 subjects in the Full Analysis Set (FAS), 502 are included in this analysis. The Last Observation Carried Forward method was utilized.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 99 | 103 | 101 | 94 | 105
Hours | 1.821 (2.655) | 2.095 (3.120) | 2.118 (2.827) | 2.364 (2.876) | 1.335 (2.975)

4. Secondary Outcome: The Change in the Relative Time Spent "on" From Baseline to the End of the Maintenance Period as Recorded by the Subject in a Daily Diary
Description: Time "On" is defined as when the patient has the effect of anti-Parkinson's medication.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 99 | 103 | 101 | 94 | 105
Hours | 12.058 (16.517) | 13.463 (20.099) | 13.410 (17.202) | 14.529 (16.531) | 9.250 (18.942)

5. Secondary Outcome: The Change in the Status of the Subject After Wake-Up From Baseline to the End of the Maintenance Period as Recorded by the Subject in a Daily Diary
Time Frame: as for outcome 1
Population: Of the 502 subjects in the Full Analysis Set (FAS), 405 are included in this analysis.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 80 | 82 | 82 | 80 | 81
Hours
  ON Without Troublesome Dyskinesias | 23.688 (41.607) | 24.593 (43.006) | 20.935 (42.132) | 21.083 (45.642) | 19.712 (41.857)
  ON With Troublesome Dyskinesias | -0.667 (18.874) | -0.813 (12.804) | 1.626 (23.659) | 1.667 (13.417) | -0.206 (8.934)
  OFF | -23.021 (40.667) | -23.780 (43.150) | -22.561 (40.519) | -22.750 (47.193) | -19.506 (43.298)

6. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part II From Baseline to the End of the Maintenance Period
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) Part II is a scale for the assessment of function in Parkinson's disease. UPDRS Part II measures Activities of Daily Living. It consists of 13 questions, each ranging from 0 to 4. The sum score of the UPDRS Part II ranges from 0 to 52. A higher score indicates greater disability. A negative change score indicates improvement.
Time Frame: as for outcome 1
Population: Of the 502 subjects in the Full Analysis Set (FAS), 497 are included in this analysis. The Last Observation Carried Forward (LOCF) method utilized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 98 | 101 | 99 | 94 | 105
units on a scale | -2.1 (4.3) | -2.2 (3.9) | -1.5 (4.7) | -2.1 (4.6) | -0.9 (3.7)

7. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part III From Baseline to the End of the Maintenance Period
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) Part III is a scale for the assessment of function in Parkinson's disease. UPDRS Part III measures Motor Function. It consists of 14 items with 27 questions, each ranging from 0 to 4. The sum score for the UPDRS Part III ranges from 0 to 108. A higher score indicates greater disability. A negative change score indicates improvement.
Time Frame: as for outcome 1
Population: Of the 502 subjects in the Full Analysis Set (FAS), 496 are included in this analysis. The Last Observation Carried Forward (LOCF) method utilized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 98 | 100 | 99 | 94 | 105
units on a scale | -3.4 (7.6) | -4.5 (7.5) | -3.5 (8.9) | -5.9 (7.6) | -2.5 (8.2)

8. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV From Baseline to the End of the Maintenance Period - What Proportion of the Waking Day Are Dyskinesias Present?
Description: Item = Duration (question #32) in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV from Baseline to the end of the Maintenance Period - What proportion of the waking day are dyskinesias present? Has a possible score of 0 - 4 points (4 = maximum). A higher score indicates more severe symptoms.
  Results show the number of subjects per dose group and their change over time either improving (decrease in score), worsening (increase in score), or remaining the same.
Time Frame: as for outcome 1
Population: Of the 502 subjects in the Full Analysis Set (FAS), 495 are included in this analysis. The Last Observation Carried Forward (LOCF) method utilized.
Measure: Number; unit: participants
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 97 | 101 | 98 | 94 | 105
participants
  Worsening | 15 | 14 | 13 | 15 | 12
  Equal | 74 | 72 | 75 | 69 | 84
  Improvement | 8 | 15 | 10 | 10 | 9

9. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV From Baseline to the End of the Maintenance Period - Disability: How Disabling Are the Dyskinesias?
Description: Item = Disability (question #33) in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV from Baseline to the end of the Maintenance Period - How disabling are the dyskinesias? Has a possible score of 0 - 4 points (4 = maximum). A higher score indicates more severe symptoms.
  Results show the number of subjects per dose group and their change over time either improving (decrease in score), worsening (increase in score), or remaining the same.
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 97 | 101 | 98 | 94 | 105
participants
  Worsening | 7 | 6 | 2 | 6 | 9
  Equal | 80 | 89 | 86 | 78 | 90
  Improvement | 10 | 6 | 10 | 10 | 6

10. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV From Baseline to the End of the Maintenance Period - Painful Dyskinesias: How Painful Are the Dyskinesias?
Description: Item = Painful Dyskinesia (question #34) in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV from Baseline to the end of the Maintenance Period - How painful are the dyskinesias? Has a possible score of 0 - 4 points (4 = maximum). A higher score indicates more severe symptoms.
  Results show the number of subjects per dose group and their change over time either improving (decrease in score), worsening (increase in score), or remaining the same.
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 97 | 101 | 98 | 94 | 105
participants
  Worsening | 2 | 3 | 4 | 2 | 8
  Equal | 90 | 94 | 86 | 87 | 94
  Improvement | 5 | 4 | 8 | 5 | 3

11. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV From Baseline to the End of the Maintenance Period - Presence of Early Morning Dystonia
Description: Item = Presence of Early Morning Dystonia (question #35) in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV from Baseline to the end of the Maintenance Period has a possible score of 0 (no) or 1 (yes). A score of 1 indicates early morning dystonia.
  Results show the number of subjects per dose group and their change over time either improving (decrease in score), worsening (increase in score), or remaining the same.
Time Frame: as for outcome 1
Population: Of the 502 subjects in the Full Analysis Set (FAS), 495 are included in this analysis. The Last Observation Carried Forward (LOCF) method was utilized.
Measure: Number; unit: participants
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 97 | 101 | 98 | 94 | 105
participants
  Worsening | 5 | 9 | 7 | 6 | 14
  Equal | 81 | 79 | 78 | 76 | 82
  Improvement | 11 | 13 | 13 | 12 | 9

12. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV From Baseline to the End of the Maintenance Period - Are "Off" Periods Predictable?
Description: Item = Are "off" periods predictable (question #36) in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV from Baseline to the end of the Maintenance Period has a possible score of 0 (no) or 1 (yes). A score of 1 indicates "off" periods are predictable.
  Results show the number of subjects per dose group and their change over time either improving (decrease in score), worsening (increase in score), or remaining the same.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 97 | 101 | 98 | 94 | 105
participants
  Worsening | 6 | 4 | 12 | 3 | 11
  Equal | 80 | 82 | 74 | 80 | 85
  Improvement | 11 | 15 | 12 | 11 | 9

13. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV From Baseline to the End of the Maintenance Period - Are "Off" Periods Unpredictable?
Description: Item = Are "off" periods unpredictable (question #37) in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV from Baseline to the end of the Maintenance Period has a possible score of 0 (no) or 1 (yes). A score of 1 indicates "off" periods are unpredictable.
  Results show the number of subjects per dose group and their change over time either improving (decrease in score), worsening (increase in score), or remaining the same.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 97 | 101 | 98 | 94 | 105
participants
  Worsening | 15 | 12 | 8 | 8 | 12
  Equal | 71 | 78 | 73 | 75 | 77
  Improvement | 11 | 11 | 17 | 11 | 16

14. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV From Baseline to the End of the Maintenance Period - Do "Off" Periods Come on Suddenly?
Description: Item = Do "off" periods come on suddenly, within a few seconds (question #38) in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV from Baseline to the end of the Maintenance Period has a possible score of 0 (no) or 1 (yes). A score of 1 indicates "off" periods come on suddenly, within a few seconds.
  Results show the number of subjects per dose group and their change over time either improving (decrease in score), worsening (increase in score), or remaining the same.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 97 | 101 | 98 | 94 | 105
participants
  Worsening | 6 | 7 | 11 | 9 | 15
  Equal | 80 | 83 | 75 | 67 | 75
  Improvement | 11 | 11 | 12 | 18 | 15

15. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV From Baseline to the End of the Maintenance Period - What Proportion of the Waking Day is the Subject "Off", on Average?
Description: Item = What proportion of the waking day is the subject "off", on average (question #39) in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV from Baseline to the end of the Maintenance Period has a possible score of 0 - 4 points (4 = maximum). A higher score indicates the subject is "off" a larger portion of the waking day.
  Results show the number of subjects per dose group and their change over time either improving (decrease in score), worsening (increase in score), or remaining the same.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 97 | 101 | 98 | 94 | 105
participants
  Worsening | 8 | 4 | 8 | 7 | 11
  Equal | 52 | 58 | 58 | 55 | 61
  Improvement | 37 | 39 | 32 | 32 | 33

16. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV From Baseline to the End of the Maintenance Period - Does the Patient Have Anorexia, Nausea, or Vomiting?
Description: Item = Does the patient have anorexia, nausea, or vomiting (question #40) in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV from Baseline to the end of the Maintenance Period has a possible score of 0 (no) or 1 (yes). A score of 1 indicates subject has anorexia, nausea, or vomiting.
  Results show the number of subjects per dose group and their change over time either improving (decrease in score), worsening (increase in score), or remaining the same.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 97 | 101 | 98 | 94 | 105
participants
  Worsening | 4 | 2 | 3 | 5 | 3
  Equal | 88 | 96 | 90 | 85 | 96
  Improvement | 5 | 3 | 5 | 4 | 6

17. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV From Baseline to the End of the Maintenance Period - Does the Patient Have Any Sleep Disturbances Such as Insomnia or Hypersomnolence?
Description: Item = Does the patient have any sleep disturbances such as insomnia or hypersomnolence (question #41) in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV from Baseline to the end of the Maintenance Period has a possible score of 0 (no) or 1 (yes). A score of 1 indicates subject has sleep disturbances such as insomnia or hypersomnolence.
  Results show the number of subjects per dose group and their change over time either improving (decrease in score), worsening (increase in score), or remaining the same.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 97 | 101 | 98 | 94 | 105
participants
  Worsening | 13 | 14 | 7 | 4 | 12
  Equal | 70 | 72 | 75 | 77 | 78
  Improvement | 14 | 15 | 16 | 13 | 15

18. Secondary Outcome: The Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV From Baseline to the End of the Maintenance Period - Does the Patient Have Symptomatic Orthostasis?
Description: Item = Does the patient have symptomatic orthostasis (question #42) in the Unified Parkinson's Disease Rating Scale (UPDRS) Part IV from Baseline to the end of the Maintenance Period has a possible score of 0 (no) or 1 (yes). A score of 1 indicates subject has symptomatic orthostasis.
  Results show the number of subjects per dose group and their change over time either improving (decrease in score), worsening (increase in score), or remaining the same.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 97 | 101 | 98 | 94 | 105
participants
  Worsening | 0 | 6 | 2 | 4 | 8
  Equal | 91 | 93 | 92 | 88 | 91
  Improvement | 6 | 2 | 4 | 2 | 6

19. Secondary Outcome: The Change in Number of "Off" Periods From Baseline to the End of the Maintenance Period as Recorded by the Subject in a Daily Diary
Description: Time "Off" is defined as when the patient does not have the effect of anti-Parkinson's medication.
Time Frame: as for outcome 1
Population: Of the 502 subjects in the Full Analysis Set (FAS), 405 are included in this analysis. The Observed Cases (OC) method was utilized.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Number analyzed (Participants) | 80 | 82 | 82 | 80 | 81
Hours | -1.144 (1.687) | -1.294 (1.971) | -1.323 (1.348) | -1.304 (1.442) | -1.006 (1.474)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected during the course of the trial, which was approximately 33 weeks per subject.
Description: Adverse Events refer to the Safety Set (SS). The Safety Set (SS) consisted of all subjects who were randomized and received at least 1 dose of study medication.
Arm/Group | Rotigotine 2 mg/24 hr | Rotigotine 4 mg/24 hr | Rotigotine 6 mg/24 hr | Rotigotine 8 mg/24 hr | Placebo
Serious Adverse Events (participants affected / at risk) | 4/101 | 3/107 | 2/104 | 0/94 | 5/108
Other Adverse Events (participants affected / at risk) | 54/101 | 54/107 | 49/104 | 52/94 | 54/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine 2 mg/24 hr (N=101) | Rotigotine 4 mg/24 hr (N=107) | Rotigotine 6 mg/24 hr (N=104) | Rotigotine 8 mg/24 hr (N=94) | Placebo (N=108)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep attacks (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine 2 mg/24 hr (N=101) | Rotigotine 4 mg/24 hr (N=107) | Rotigotine 6 mg/24 hr (N=104) | Rotigotine 8 mg/24 hr (N=94) | Placebo (N=108)
Nausea (Gastrointestinal disorders) | 13 (17) | 11 (12) | 15 (19) | 11 (11) | 8 (10)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 8 (8) | 4 (5) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 7 (8) | 7 (7) | 5 (5) | 0 (0)
Fatigue (General disorders) | 7 (7) | 5 (5) | 2 (2) | 4 (4) | 6 (7)
Application site pruritus (General disorders) | 4 (4) | 6 (6) | 8 (8) | 7 (8) | 2 (2)
Application site erythema (General disorders) | 4 (4) | 5 (5) | 7 (8) | 5 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (8) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 6 (6) | 0 (0) | 2 (2) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 7 (9) | 6 (7) | 4 (12) | 6 (6) | 7 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 5 (5) | 5 (6) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 3 (3) | 5 (8) | 3 (3)
Headache (Nervous system disorders) | 10 (11) | 8 (8) | 6 (7) | 8 (10) | 12 (18)
Dizziness (Nervous system disorders) | 8 (8) | 11 (12) | 7 (9) | 6 (6) | 9 (9)
Somnolence (Nervous system disorders) | 7 (8) | 6 (6) | 8 (11) | 4 (4) | 9 (10)
Dyskinesia (Nervous system disorders) | 5 (6) | 4 (4) | 11 (11) | 14 (18) | 3 (6)
Tremor (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3) | 5 (5) | 3 (7)
Insomnia (Psychiatric disorders) | 6 (6) | 8 (9) | 6 (6) | 6 (6) | 7 (8)
Confusional state (Psychiatric disorders) | 5 (5) | 2 (2) | 6 (6) | 1 (1) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.